CLINICAL TRIAL: NCT04616495
Title: Liver Transplantation in Patients With Unresectable Colorectal Liver Metastases
Acronym: TRASMETIR
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Eva M. Montalvá, Hepatobiliarypancreatic and Transplant Surgeon, Hospital Universitario La Fe
Other Study IDs: TRASMETIR
Record Dates: First submitted 2020-09-25; First posted 2020-11-05 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer; Metastatic Liver Cancer; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver transplanted patients
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation — Chemotherapy and liver transplantation

SUMMARY:
Multicentric prospective and observational study to assess the 5-year overall survival in a cohort of patients with unresectable liver-only colorectal metastases, well controlled by chemotherapy prior to liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ years
* Good performance status, ECOG 0 or 1
* Resected adenocarcinoma in colon or rectum (R0 resection)
* Unresectable liver metastases
* No extrahepatic disease
* Normal blood tests
* Response to ≤ 2 lines of chemotherapy (RECIST criteria)
* ≥ 1 year period since diagnosis of colorectal cancer to enrolment in liver transplant waiting list
* Signed informed consent

Exclusion Criteria:

* Body mass index ≥ 30
* Positive HIV or HCV
* Pregnancy at the time of inclusion
* BRAF mutated status
* Deterioration of general condition (10% weight loss in the prior 6 months)
* Other malignancy with disease free survival < 5 years
* Concomitant or prior extrahepatic metastases (histologically or radiologically proved), even if surgically resected.
* Palliative resection of primary colorectal adenocarcinoma
* Liver metastases size > 5 cm (in the last imaging technique)
* CEA > 80 ng/ml (at time of enrolment in waiting list)
* No neoadjuvant chemotherapy treatment
* General contraindication to liver transplantation

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cohort of patients detected in oncological units where they have been treated for colorectal cancer (stage IV with liver only unresectable metastases)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
five year overall survival (OS) | 5 years

SECONDARY OUTCOMES:
one year disease free survival (DFS) | 1 year
three year disease free survival (DFS) | 3 years
five year disease free survival (DFS) | 5 years
Quality of life using EORTC questionnaires: QLQ-C30 | 1 year
Quality of life using EORTC questionnaires: QLQ-C30 | 3 years
Quality of life using EORTC questionnaires: QLQ-C30 | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Eva M Montalvá, Valencia, Spain